CLINICAL TRIAL: NCT00188162
Title: Can Minimum Dose CT Post Lung Biopsy Predict Patient Outcome?
Brief Title: Minimum Dose CT Post Lung Biopsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 03-0898
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2007-04-23 (Estimated); Status verified 2005-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

INTERVENTIONS:
Device: CT

SUMMARY:
The aim is to evaluate whether Minimum Dose CT (MnDCT) is useful in the management of patients post Lung Biopsy

DETAILED DESCRIPTION:
Patients post Lung Biopsy have a chest X-ray (CXR) and a MnDCT post lung biopsy. Both studies are compared for the detection of a pneumothorax

ELIGIBILITY:
Inclusion Criteria:

* All Patients having a lung biopsy

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2004-01; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Detection of Pneumothorax

CONTACTS AND LOCATIONS:
Overall Officials: Narinder Paul, FRCP C, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada